CLINICAL TRIAL: NCT04674657
Title: Does Extra-Corporeal Membrane Oxygenation Alter Anti-infectives Therapy Pharmacokinetics in Adult Critically Ill Patients
Brief Title: Does Extra-Corporeal Membrane Oxygenation Alter Antiinfectives Therapy Pharmacokinetics in Critically Ill Patients
Acronym: EAT-PK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18/LO/0691
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Critical Illness; Extracorporeal Membrane Oxygenation Complication; Infection
MeSH Terms: conditions — Critical Illness; Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- caspofungin: Adult critically ill patients on ECMO receiving caspofungin therapy
  Interventions: Drug: blood drug concentration
- posaconazole: Adult critically ill patients on ECMO receiving posaconazole therapy
  Interventions: Drug: blood drug concentration

INTERVENTIONS:
Drug: blood drug concentration — blood drug concentration

SUMMARY:
Observational study Primary Objective: To study whether ECMO alters the PK of anti-infectives including voriconazole, posaconazole and caspofungin in critically ill patients on ECMO

Secondary Objectives:

Develop Population PK models of anti-infectives, including voriconazole, posaconazole and caspofungin in critically ill patients on ECMO

Develop Physiological-Based PK (PBPK) model of anti-infectives, including: voriconazole, posaconazole and caspofungin in critically ill patients on ECMO

Study population: Critically ill patients on ECMO

Methodology: Observational study to determine whether ECMO alters the PK of anti-infectives, by developing PK models

This is a non-interventional descriptive study in that the anti-infective drug selection and dosing will be at the discretion of the clinician, based on the clinical context and unit guidelines. Doses will be reconstituted and administered as per local hospital protocols in line with patient's routine care. Patients will be asked to provide additional blood samples over the course of the anti-infective dosing schedule, these samples will be taken from existing arterial lines to help guide treatment in future patients on ECMO receiving these anti-infectives.

DETAILED DESCRIPTION:
Anti-infective drug selection and dosing will be at the discretion of the clinician, based on the clinical context and unit guidelines. Doses will be reconstituted and administered as per local hospital protocols and based on routine standard care.

Blood samples will be drawn from an existing arterial line and collected in 3 ml tubes with Lithium Heparin anticoagulant.

All patients will be sampled over a single dosing period on the second day of Extra-Corporeal Membrane Oxygenation (ECMO) treatment, or of an antibiotic course where antibiotics are commenced whilst the patient is on ECMO. Where possible, sampling during one extra dosing interval will occur on days 4-8 of ECMO treatment and/or prior to the next tubing change. Where two or more anti-infectives of interest are prescribed for one patient, collect data on timing of administration for both drugs and sample according to the antibiotic with the longer dosing interval.

Blood samples (2ml) will be collected from an existing arterial line at the following time points 0 (pre-starting infusion, pre-Nasogastric (NG)/Oral (PO) dose), 1 (end of infusion or 1hour post NG/PO dose), 2, 3, 4, 8 and either 12 (for twice daily regimen) or 24 (for once daily regimen) hours on the second day of ECMO.

Where a patient is receiving medications where a validated drug assay exists in addition to the study drug (such as other anti-infectives), analysis of the additional therapy will also be attempted where practical.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years and <90 years
2. Currently undergoing ECMO for respiratory +/- cardiac dysfunction
3. Clinical indication for the anti-infectives, including voriconazole, posaconazole and caspofungin

Exclusion Criteria:

1. History of allergy to any of the study drug
2. Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients on Extra-Corporeal Membrane Oxygenation
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-09-03 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve (AUC) of Caspofungin in adult critically ill patients on ECMO | 24 hour
  Blood samples (2ml) will be collected from an existing arterial line at the following time points 0 (pre-starting infusion, pre-NG/PO dose), 1 (end of infusion or 1hour post NG/PO dose), 2, 3, 4, 8 and either 12 (for twice daily regimen) or 24 (for once daily regimen) hours on the second day of ECMO
Area Under the Plasma Concentration Versus Time Curve (AUC) of Posaconazole in adult critically ill patients on ECMO | 24 hour
  Blood samples (2ml) will be collected from an existing arterial line at the following time points 0 (pre-starting infusion, pre-NG/PO dose), 1 (end of infusion or 1hour post NG/PO dose), 2, 3, 4, 8 and either 12 (for twice daily regimen) or 24 (for once daily regimen) hours on the second day of ECMO

CONTACTS AND LOCATIONS:
Overall Officials: Anna Reed, Principal Investigator — Royal Brompton and Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton & Harefield NHS Foundation Trust, Harefield, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT04674657/Prot_SAP_000.pdf